CLINICAL TRIAL: NCT02474719
Title: Transfer and Ultrafiltration In Peritoneal Dialysis
Acronym: TULIPE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: few eligible patients, dialysate drainage problem, measurement bias : not all currently marketed laboratory instruments are able to dose peritoneal dialysate
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TULIPE
Record Dates: First submitted 2015-06-03; First posted 2015-06-18 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2017-02

CONDITIONS: End-stage Renal Disease
Keywords: nephrology; extra-renal purification; peritoneal dialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Peritoneal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional scheme followed by alternate schem (Experimental): The first day of the study, patients receive an adapted conventional peritoneal dialysis scheme: 2 cycles of ultrafiltration (stasis: 35 mn ; volume: 650cc/m²) and 2 cycles of purification (stasis: 110 mn ; volume 1200cc/m²).
  The second day, patients receive an adapted and alternate scheme: 1 cycle of ultrafiltration (stasis: 35 mn ; volume: 650cc/m²) and 1 cycle of purification (stasis: 110 mn ; volume 1200cc/m²), the two cycles being repeated once.
  Interventions: Other: comparison of two regimens in peritoneal dialysis
- alternate scheme followed by conventional scheme (Experimental): The first day of the study, patients receive an adapted and alternate peritoneal dialysis scheme: 1 cycle of ultrafiltration (stasis: 35 mn ; volume: 650cc/m²) and 1 cycle of purification (stasis: 110 mn ; volume 1200cc/m²), the two cycles being repeated once.
  The second day, patients receive an adapted conventional scheme: 2 cycles of ultrafiltration (stasis: 35 mn ; volume: 650cc/m²) and 2 cycles of purification (stasis: 110 mn ; volume 1200cc/m²).
  Interventions: Other: comparison of two regimens in peritoneal dialysis

INTERVENTIONS:
Other: comparison of two regimens in peritoneal dialysis — Dialysate samples (8 by scheme, volume of 10 mL) are collected at each cycle (one at the beginning and one at the end of the cycle). A blood sample (5 mL) is collected at the beginning of the second scheme and a 24-hour urine sample at the end of the second scheme.

SUMMARY:
The aim of this study is to demonstrate the efficiency of an adapted and "alternate" peritoneal dialysis scheme in terms of sodium extraction and purification compared to an adapted conventional peritoneal dialysis scheme.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in the Nephrology department of the Besançon University Hospital
* Patients treated by continuous ambulatory peritoneal dialysis or ambulatory peritoneal dialysis for at least 6 months
* Absence of hospitalization caused by an infection in the month prior to inclusion
* Patients with a ratio (D / P) of the concentration of creatinine in the blood and dialysate between 0.5 and 0.8 on a checkup of less than 1 year.
* No contraindication to the use of hypertonic bag
* Signature of informed consent for participation indicating that the subject has understood the purpose and procedures required by the study and agrees to participate in the study and comply with the requirements and limitations inherent in this study
* Affiliation to a French social security system or beneficiary

Exclusion Criteria:

* Legal incapacity or limited legal capacity
* Patients unlikely to cooperate in the study and/or low cooperation anticipated by the investigator
* Patients without health insurance
* Pregnant women
* Patient being in the exclusion period from another study or planned by the "national register of volunteers"
* Hospitalization caused by an infection in the month prior to inclusion
* Patients with a peritoneal dialysis catheter dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-01; Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Intra-dialytic concentrations of different electrolytes (sodium, phosphorus, urea, creatinine, glucose and proteins) | In a maximum of 72 hours after collection

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Courivaud, MCU/PH, Principal Investigator — Besançon University Hospital, nephrology department
Locations (1):
- Besançon University Hospital, Nephrology Department, Besançon, Franche-Comté, France